CLINICAL TRIAL: NCT02199938
Title: Identification and Characterization of Molecular Markers in Musculoskeletal Tumors
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator has left the Institution
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EK 10/2007 (5)
Record Dates: First submitted 2014-07-01; First posted 2014-07-25 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Soft Tissue and Bone Tumors; Sarcoma; Sarcoma of Bone; Soft Tissue Sarcoma
MeSH Terms: conditions — Bone Neoplasms; Sarcoma; Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood serum blood plasma tumor tissue tumor free tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- musculoskeletal tumors: Patients with suspected or confirmed bone or soft tissue tumors undergoing biopsy or surgery
  Interventions: Other: Identification and characterization of molecular markers in musculoskeletal tumors

INTERVENTIONS:
Other: Identification and characterization of molecular markers in musculoskeletal tumors

SUMMARY:
The aim of the study is to improve the understanding of molecular mechanisms in the development and progression of musculoskeletal tumors. These tumors do have in general unfavorable prognosis and conventional treatments (e.g. surgery, radiotherapy or chemotherapy) could not enhance the prognosis of these patients during the last ten to fifteen years. Therefore the investigators chose a new way, as they try to identify markers on a genetic level, who ideally act as a basis to develop new treatment options.

DETAILED DESCRIPTION:
To definitely asses such molecular markers in musculoskeletal tumors they have to be identified in human patient samples with corresponding tumors, before molecular markers can be validated in animal models. Just because these soft tissue and bone tumors are rare (compared to breast and lung carcinomas), it is of great importance that samples from all patients treated at Balgrist University Hospital are collected systematically und stored correspondingly. Only like this valid statements can be done. Therefore the investigators intent to collect tissue and blood samples from all patients who agree in participating in the study. The samples will be taken during routine biopsies and operations. To compare tumor tissue and healthy tissue it is also planed to take samples from tumor free patients who undergo a knee replacement surgery. The investigators would store the surgical waste and involve these samples in the analyzes.

Clinical data regarding diagnosis and examination findings, as well as tissue from biopsies and surgeries will be collected prospectively. The tissue will be frozen in liquid nitrogen according to standard procedures and stored until the molecular analyzes at the Laboratory of Orthopedic Research at Balgrist University Hospital. The processing involves expression analyzes such as polymerase chain reaction, Western Blot, micro arrays, immunohistochemistry and tissue array. The DNA from the taken blood samples shall be compared with the DNA found in the tumor.

ELIGIBILITY:
Inclusion Criteria:

* surgery or biopsy of a bone- or soft tissue tumor
* informed consent

Exclusion Criteria:

* patients wish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who receive a biopsy or surgery because of confirmed or suspected musculoskeletal tumor.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Tumor RNA in resected tissue | at time of surgery

SECONDARY OUTCOMES:
Cell free tumor RNA in blood plasma | 7 to 1 day before surgery
Cell free tumor RNA in blood plasma | 1 day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided